CLINICAL TRIAL: NCT03301038
Title: Rifampin to Reduce Elevated Levels of Blood and Urine Calcium in Patients With Inactivating Mutations in the CYP24A1 Gene
Brief Title: Rifampin in CYP24A1-related Hypercalcemia and Hypercalciuria
Acronym: RICHH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-013429; R01DK112955 (NIH)
Record Dates: First submitted 2017-09-01; First posted 2017-10-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Infantile Hypercalcaemia - Severe Form; Genetic Disease; Hypercalcemia, Idiopathic, of Infancy; Hypercalciuric Hypercalcemia; Idiopathic Infantile Hypercalcemia - Mild Form; Hypercalciuria
Keywords: hypercalcemia; nephrocalcinosis; CYP24A1; hypercalciuria
MeSH Terms: conditions — Genetic Diseases, Inborn; Hypercalcemia, Idiopathic, of Infancy; Hypercalciuric Hypercalcemia; Hypercalciuria; Hypercalcemia; Nephrocalcinosis | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Subjects (Experimental): SingleArm: Escalating doses of rifampin (5 and 10 mg/kg/day) (SingleArm)
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Rifampin — Rifampin 5 mg/kg (max 300 mg) daily for 8 weeks, followed by rifampin 10 mg/kg (max 600 mg) daily for 8 weeks.
  Other Names: Rifadin; Rifampicin

SUMMARY:
This study evaluates the efficacy of rifampin in the treatment of hypercalcemia and/or hypercalciuria in participants with at least one inactivating mutation of the CYP24A1 gene. Eligible subjects will receive rifampin for a total of 16 weeks during this study.

DETAILED DESCRIPTION:
Idiopathic infantile hypercalcemia (IIH; omim 143880) is a genetic disorder of mineral metabolism characterized by severe hypercalcemia and/or hypercalciuria, suppressed serum levels of parathyroid hormone (PTH) and elevated levels of the active vitamin D metabolite, 1,25(OH)2D. Biallelic inactivating mutations of CYP24A1, the gene encoding the 24-hydroxylase enzyme that represents the principal pathway for inactivation of vitamin D metabolites, cause the most common and severe form of IIH.

Investigators have preliminary data supporting a novel therapeutic approach to repurpose rifampin as an agent to induce over-expression of CYP3A4 and CYP3A5, enzymes that are expressed in the liver and intestine. When these enzymes are induced, the increased enzyme activity provides an alternative catabolic pathway for inactivation of vitamin D metabolites. The purpose of this study is to obtain support for an open label, escalating dose study to assess the effect, safety, and tolerability of once daily oral rifampin in participants with IIH due to inactivating mutations in CYP24A1.

In this study, Investigators will recruit 60 patients with at least one inactivating mutation of CYP24A1. Participants will be observed for 8-weeks before a 16-week treatment phase of rifampin and 8 further weeks of observation. In addition to following the effect of treatment on calcium homeostasis, Investigators will also study the pharmacokinetics of rifampin in this condition and the effect on intestinal calcium absorption.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 6 months to 65 years.
* at least one mutations of CYP24A1
* Serum and/or urinary calcium above the normal reference range for age
* Serum PTH concentration <20 pg/ml
* Elevated or normal serum concentration of 1,25-dihydroxyvitamin D3.

Exclusion Criteria:

* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
* Allergy to rifampin or related medications
* Current therapies with medications that have significant drug-drug interactions with rifampin, defined as a medication considered to interact with CYP3A4 or CYP3A5 and either induce or inhibit expression or function of these P450 enzymes. By "drug-drug" interactions we are looking for medications that will affect metabolism or action of rifampin as exclusionary, not medications that will be affected by rifampin.
* Pregnancy or breastfeeding
* Laboratory abnormalities that indicate clinically significant hepatic, or renal disease:
* Aspartate Aminotransferase (AST/SGOT) > 2.0 times the upper limit of normal Alanine aminotransferase (ALT/SGPT) > 2.0 times the upper limit of normal Total bilirubin > 2.0 times the upper limit of normal Creatinine > 2.0 times the upper limit of normal

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Serum albumin-adjusted calcium | up to 32 weeks
  Measured at baseline and every 4 weeks
Serum parathyroid hormone | up to 32 weeks
  Measured at baseline and every 4 weeks
Urinary calcium excretion | up to 32 weeks
  Measured at baseline and every 4 weeks

SECONDARY OUTCOMES:
Intestinal calcium absorption | baseline, 8, 16, 24 and 32 weeks post-dose
  Measured using stable calcium isotopes five times during the study
Nephrocalcinosis | Baseline and week 32
  Renal ultrasound performed before and after treatment
Rifampin pharmacokinetics | 8, 16 and 24 weeks post-dose
  Measured three times during the study

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Levine, MD, Principal Investigator — Children'sHospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hawkes CP, Li D, Hakonarson H, Meyers KE, Thummel KE, Levine MA. CYP3A4 Induction by Rifampin: An Alternative Pathway for Vitamin D Inactivation in Patients With CYP24A1 Mutations. J Clin Endocrinol Metab. 2017 May 1;102(5):1440-1446. doi: 10.1210/jc.2016-4048. PMID 28324001
- [Background] Dauber A, Nguyen TT, Sochett E, Cole DE, Horst R, Abrams SA, Carpenter TO, Hirschhorn JN. Genetic defect in CYP24A1, the vitamin D 24-hydroxylase gene, in a patient with severe infantile hypercalcemia. J Clin Endocrinol Metab. 2012 Feb;97(2):E268-74. doi: 10.1210/jc.2011-1972. Epub 2011 Nov 23. PMID 22112808
- [Background] Schlingmann KP, Kaufmann M, Weber S, Irwin A, Goos C, John U, Misselwitz J, Klaus G, Kuwertz-Broking E, Fehrenbach H, Wingen AM, Guran T, Hoenderop JG, Bindels RJ, Prosser DE, Jones G, Konrad M. Mutations in CYP24A1 and idiopathic infantile hypercalcemia. N Engl J Med. 2011 Aug 4;365(5):410-21. doi: 10.1056/NEJMoa1103864. Epub 2011 Jun 15. PMID 21675912